CLINICAL TRIAL: NCT06001034
Title: A 9-week Program of Supervised Occlusive Aerobic Training in People With Fibromyalgia in a Hospital Setting, and Its Impact on Blood/Plasma Variables, Quality of Life and Functional Autonomy.
Brief Title: Program of Supervised Occlusive Aerobic Training in People With Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Carlos Rodríguez Bautista (Other)
Collaborators: Universidad Pablo de Olavide (Other); Hospital Universitario de Valme (Other); Andaluz Health Service (Other Government)
Responsible Party: Sponsor-Investigator, José Carlos Rodríguez Bautista, PhD currently Sport Sciences in Physical Activity, Health and Quality of Life, Universidad Pablo de Olavide
Organization: Universidad Pablo de Olavide (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1441-23; 0560-N-22 (Other: PEIBA. Junta de Andalucía. Government of Spain.)
Record Dates: First submitted 2023-07-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Fibromyalgia
Keywords: occlusive training
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Group 1: Aerobic exercise plus occlusive tool. Group 2: Aerobic exercise without occlusive tool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Aerobic exercise plus occlusive tool. (Experimental): Performing low-impact aerobic exercise with an occlusive tool 2 days per week.
  Interventions: Device: Occlusion training
- Group 2: Aerobic exercise without occlusive tool. (No Intervention): Performing low-impact aerobic exercise without an occlusive tool 2 days per week.

INTERVENTIONS:
Device: Occlusion training — Impact of supervised occlusive training for 2 days per week for 10 weeks on quality of life and functional autonomy in participants with fibromyalgia.
  Other Names: Occlusive cuffing during aerobic exercise in participants with fibromyalgia
  Arms: Group 1: Aerobic exercise plus occlusive tool.

SUMMARY:
Occlusive training in people with fibromyalgia

DETAILED DESCRIPTION:
Intervention study in people with fibromyalgia with the implementation of a lower body occlusive tool in aerobic exercise. The study aims to descriptively test the impact on quality of life and functional autonomy of occlusive training in a controlled and individualized way in two groups: group 1 aerobic exercise with use of occlusive tool and group 2, aerobic exercise without occlusive tool in a period of 9 weeks twice a week.

ELIGIBILITY:
Inclusion Criteria:

A patient meets diagnostic criteria for fibromyalgia if the following three conditions are present: (American Rheumatology Association). Wolfe et al., (2010).

* o 1) Widespread Pain Index (WPI) ≥ 7 and Symptom Severity Score (SS Score) ≥ 5 or WPI 3-6 and SS ≥ 9.
* Symptoms have been present, at a similar level, during the last three months.
* The patient has no other pathology that could explain the pain.
* Recent negative COVID-19 test.

Exclusion Criteria:

* Other associated pathologies that may hinder the development of the research.
* Mobility limitations.
* Injuries that add to those of the disease itself and hinder mobility.
* No medical evaluation of the diagnosis of the disease.
* Negative results in the inclusion tests.
* Cardiac pathologies.
* Blood pressure higher than 130-90 mmHg.
* No COVID-19 test.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Coenzyme Q10 after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  Coenzyme Q10
Change in total antioxidants after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  TAS
Change in disease impact questionnaire WPI after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  WPI; score between (0-19). The higher the score, the greater the impact of the disease.
Change in disease impact questionnaire SSscore after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  SS score; score between (0-3) in the first half. Score between (0-40); between 1-10 (1 point), between 11-24 (2 points), more than 25 (3 points) in the second half. The higher the score, the greater the impact of the disease.
Change in disease impact questionnaire FIQ after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  FIQ; score between (0-100). The higher the score, the greater the impact of the disease
Change in disease impact questionnaire MFI-20 after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  MFI-20; (0-60) no fatigue. (60-70), fatigue, lighter or more severe, depending on the depending on the rating closer to 60 or 70 points. (more than 70 points), severe fatigue.
Change in high density lipoproteins after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  HDL
Change in low density lipoproteins after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  LDL
Change in total cholesterol lipoproteins after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  CHOL
Change in triglycerides after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  TG
Changes in urea after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  Urea
Changes in creatinine after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  Creatinine
Change in gamma-glutamyl transferase after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  GGT
Change in glutamic-pyruvic transaminase after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  GPT
Change in glutamic oxaloacetic acid transaminase after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  GOT
Change in alkaline phosphatase after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  ALP
Change in funcional test after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period)
  6-minute walking test
Change in funcional test after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period)
  incremental shuttle walking test
Change in funcional test after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  30 second chair and stand test
Change in funcional test after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period)
  Time and go test
Change in malondialdehyde after a 9-week intervention period. | Pre (before the start of the 9-week intervention period). Post (immediately after the 9-week intervention period).
  MDA (malondialdehyde)
Change in distance traveled after a 9-week intervention period. | From week 1 to week 9 of the intervention period.
  Pedometer registration. Immediately after each session from week 1 to 9 of the intervention period. With a total of 18 recordings over the 9 weeks of the intervention period.
Change in visual pain scale VAS over a 9-week intervention period. | From week 1 to week 9 of the intervention period.
  Visual pain scale (1-10). 1 being lighter and 10 being more severe. Visual pain scale recording. Before and immediately after each session from week 1 to week 9 of the intervention period. With a total of 36 recordings during the 9 weeks of the intervention period.
Change in perceived exertion scale BORG over a 9-week intervention period. | From week 1 to week 9 of the intervention period.
  Perceived exertion scale. (1-10). 1 being lighter and 10 being more severe. Perceived exertion scale recording. Before and immediately after each session from week 1 to week 9 of the intervention period. With a total of 36 recordings during the 9 weeks of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Rodríguez Bautista, PhD currently, Principal Investigator — Universidad Pablo de Olavide
Locations (1):
- Universidad Pablo de Olavide, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Numeric code to each participant, concealing their personal data at all times.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The protocol before the start and the numerical codes at the end of the intervention period.
Access Criteria: Shared use only from principal investigator with collaborating investigators of the study.

REFERENCES:
- [Background] Latorre-Roman PA, Segura-Jimenez V, Aparicio VA, Santos E Campos MA, Garcia-Pinillos F, Herrador-Colmenero M, Alvarez-Gallardo IC, Delgado-Fernandez M. Ageing influence in the evolution of strength and muscle mass in women with fibromyalgia: the al-Andalus project. Rheumatol Int. 2015 Jul;35(7):1243-50. doi: 10.1007/s00296-015-3213-5. Epub 2015 Jan 24. PMID 25617055
- [Background] Bonaterra GA, Then H, Oezel L, Schwarzbach H, Ocker M, Thieme K, Di Fazio P, Kinscherf R. Morphological Alterations in Gastrocnemius and Soleus Muscles in Male and Female Mice in a Fibromyalgia Model. PLoS One. 2016 Mar 17;11(3):e0151116. doi: 10.1371/journal.pone.0151116. eCollection 2016. PMID 26986947
- [Background] Valim V, Oliveira LM, Suda AL, Silva LE, Faro M, Neto TL, Feldman D, Natour J. Peak oxygen uptake and ventilatory anaerobic threshold in fibromyalgia. J Rheumatol. 2002 Feb;29(2):353-7. PMID 11842825
- [Background] Koca I, Savas E, Ozturk ZA, Boyaci A, Tutoglu A, Alkan S, Yildiz H, Kimyon G. The evaluation in terms of sarcopenia of patients with fibromyalgia syndrome. Wien Klin Wochenschr. 2016 Nov;128(21-22):816-821. doi: 10.1007/s00508-015-0821-8. Epub 2015 Jul 4. PMID 26142171
- [Background] Shang Y, Gurley K, Symons B, Long D, Srikuea R, Crofford LJ, Peterson CA, Yu G. Noninvasive optical characterization of muscle blood flow, oxygenation, and metabolism in women with fibromyalgia. Arthritis Res Ther. 2012 Nov 1;14(6):R236. doi: 10.1186/ar4079. PMID 23116302
- [Background] Sarifakioglu B, Guzelant AY, Guzel EC, Guzel S, Kiziler AR. Effects of 12-week combined exercise therapy on oxidative stress in female fibromyalgia patients. Rheumatol Int. 2014 Oct;34(10):1361-7. doi: 10.1007/s00296-014-2978-2. Epub 2014 Mar 9. PMID 24610539
- [Background] Cordero MD, de Miguel M, Moreno-Fernandez AM. [Mitochondrial dysfunction in fibromyalgia and its implication in the pathogenesis of disease]. Med Clin (Barc). 2011 Mar 12;136(6):252-6. doi: 10.1016/j.medcli.2010.01.030. Epub 2010 Apr 24. Spanish. PMID 20417529
- [Background] Sprott H, Salemi S, Gay RE, Bradley LA, Alarcon GS, Oh SJ, Michel BA, Gay S. Increased DNA fragmentation and ultrastructural changes in fibromyalgic muscle fibres. Ann Rheum Dis. 2004 Mar;63(3):245-51. doi: 10.1136/ard.2002.004762. PMID 14962957
- [Background] Castro-Marrero J, Cordero MD, Saez-Francas N, Jimenez-Gutierrez C, Aguilar-Montilla FJ, Aliste L, Alegre-Martin J. Could mitochondrial dysfunction be a differentiating marker between chronic fatigue syndrome and fibromyalgia? Antioxid Redox Signal. 2013 Nov 20;19(15):1855-60. doi: 10.1089/ars.2013.5346. Epub 2013 May 29. PMID 23600892
- [Background] Emerling BM, Weinberg F, Snyder C, Burgess Z, Mutlu GM, Viollet B, Budinger GR, Chandel NS. Hypoxic activation of AMPK is dependent on mitochondrial ROS but independent of an increase in AMP/ATP ratio. Free Radic Biol Med. 2009 May 15;46(10):1386-91. doi: 10.1016/j.freeradbiomed.2009.02.019. Epub 2009 Mar 3. PMID 19268526
- [Background] Laderoute KR, Amin K, Calaoagan JM, Knapp M, Le T, Orduna J, Foretz M, Viollet B. 5'-AMP-activated protein kinase (AMPK) is induced by low-oxygen and glucose deprivation conditions found in solid-tumor microenvironments. Mol Cell Biol. 2006 Jul;26(14):5336-47. doi: 10.1128/MCB.00166-06. PMID 16809770
- [Background] Collado-Mateo D, Dominguez-Munoz FJ, Adsuar JC, Merellano-Navarro E, Olivares PR, Gusi N. Reliability of the Timed Up and Go Test in Fibromyalgia. Rehabil Nurs. 2018 Jan/Feb;43(1):35-39. doi: 10.1002/rnj.307. PMID 27781288
- [Background] Heredia-Jimenez J, Latorre-Roman P, Santos-Campos M, Orantes-Gonzalez E, Soto-Hermoso VM. Spatio-temporal gait disorder and gait fatigue index in a six-minute walk test in women with fibromyalgia. Clin Biomech (Bristol). 2016 Mar;33:1-6. doi: 10.1016/j.clinbiomech.2016.01.009. Epub 2016 Feb 2. PMID 26878719
- [Background] Pankoff BA, Overend TJ, Lucy SD, White KP. Reliability of the six-minute walk test in people with fibromyalgia. Arthritis Care Res. 2000 Oct;13(5):291-5. doi: 10.1002/1529-0131(200010)13:53.0.co;2-x. PMID 14635298
- [Background] Salvi D, Poffley E, Orchard E, Tarassenko L. The Mobile-Based 6-Minute Walk Test: Usability Study and Algorithm Development and Validation. JMIR Mhealth Uhealth. 2020 Jan 3;8(1):e13756. doi: 10.2196/13756. PMID 31899457
- [Background] Wevers LE, Kwakkel G, van de Port IG. Is outdoor use of the six-minute walk test with a global positioning system in stroke patients' own neighbourhoods reproducible and valid? J Rehabil Med. 2011 Nov;43(11):1027-31. doi: 10.2340/16501977-0881. PMID 22031349
- [Background] Southard V, Gallagher R. The 6MWT: will different methods of instruction and measurement affect performance of healthy aging and older adults? J Geriatr Phys Ther. 2013 Apr-Jun;36(2):68-73. doi: 10.1519/JPT.0b013e318264b5e8. PMID 22871787
- [Background] Burr JF, Bredin SS, Faktor MD, Warburton DE. The 6-minute walk test as a predictor of objectively measured aerobic fitness in healthy working-aged adults. Phys Sportsmed. 2011 May;39(2):133-9. doi: 10.3810/psm.2011.05.1904. PMID 21673494
- [Background] Ratter J, Radlinger L, Lucas C. Several submaximal exercise tests are reliable, valid and acceptable in people with chronic pain, fibromyalgia or chronic fatigue: a systematic review. J Physiother. 2014 Sep;60(3):144-50. doi: 10.1016/j.jphys.2014.06.011. Epub 2014 Jul 30. PMID 25084634
- [Background] Leone M, Duverge S, Kalinova E, Bui HT, Comtois AS. Comparison of bioenergetics of walking during a multistage incremental shuttle walk test and a 6-min walk test in active older adults. Aging Clin Exp Res. 2017 Apr;29(2):239-246. doi: 10.1007/s40520-016-0555-0. Epub 2016 Mar 14. PMID 26971801
- See also: 30-second chair stand — https://upotv.upo.es/video/58da21db238583e0478b48f3
- See also: Timed Up and Go test — https://www.youtube.com/watch?v=8eRQexJzzUE
- See also: 6-Minute Walk test — https://upotv.upo.es/video/5936500f238583f9658b464a
- See also: Incremental Shuttle Walk Test — https://upotv.upo.es/video/5a72df02238583bd408b456a

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT06001034/Prot_SAP_000.pdf